CLINICAL TRIAL: NCT01502007
Title: Activity Monitoring and Counseling in a Geriatric Population: a Randomized Trial
Brief Title: Activity Monitoring and Counseling in a Geriatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: JR Albert Foundation (Unknown)
Responsible Party: Principal Investigator, Warren G. Thompson, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-008672
Record Dates: First submitted 2011-11-29; First posted 2011-12-30 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Overweight; Obesity
Keywords: Activity Level; Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accelerometer feedback and lifestyle counseling (Experimental): The accelerometer, Fitbit, will be worn continuously. Fitbit can provide feedback to subjects about their physical activity. Subjects will wear the Fitbit for two weeks (without feedback) to obtain baseline activity data. The experimental group will then be instructed on use of the fitbit. Subjects will meet with the exercise counselor who will use accelerometer data to provide feedback and counseling to help the user increase their activity by at least 20% each day. In subjects who achieve an increase of 20%, the counseling will focus either on maintaining activity levels or increasing activity further depending on the desire of the subject. Counseling will be provided once weekly by phone and in person at least once a month. Following the 26th week the experimental subjects will continue to wear the Fitbit and receive feedback about their activity levels for an additional 24 weeks, but they will no longer receive counseling.
  Interventions: Other: Accelerometer feedback and lifestyle counseling
- Accelerometer without Feedback (Experimental): The accelerometer, Fitbit, will be worn continuously. Subjects will wear the Fitbit for two weeks (without feedback) to obtain baseline activity data. The control group will continue to wear the fitbit for the next 24 weeks without any feedback or activity counseling. Following the 26th week of the study, the subjects in the control group will complete the same program given to the experimental group in weeks 2 through 26.
  Interventions: Other: Accelerometer without Feedback

INTERVENTIONS:
Other: Accelerometer feedback and lifestyle counseling — Subjects will meet with the exercise counselor who will use accelerometer data to provide feedback and counseling to help the user increase their activity by at least 20% each day. In subjects who achieve an increase of 20%, the counseling will focus either on maintaining activity levels or increasing activity further depending on the desire of the subject. Counseling will be provided once weekly by phone and in person at least once a month. Following the 26th week the experimental subjects will continue to wear the Fitbit and receive feedback about their activity levels for an additional 24 weeks, but they will no longer receive counseling. The control group will receive no counseling for the first 26 weeks of the study and will then crossover to get accelerometry feedback and counseling for the last 24 weeks of the study.
  Arms: Accelerometer feedback and lifestyle counseling
Other: Accelerometer without Feedback — The accelerometer, Fitbit, will be worn continuously. Fitbit can provide feedback to subjects about their physical activity. Subjects will wear the Fitbit for two weeks (without feedback) to obtain baseline activity data. The experimental group will then be instructed on use of the fitbit. This group will receive feedback from the accelerometer for the remainder of the study. The control group will wear the Fitbit but receive no feedback for the first 26 weeks of the study. For the last 24 weeks they will crossover and receive feedback from the Fitbit accelerometer.
  Arms: Accelerometer without Feedback

SUMMARY:
The goal of the study is to determine if a Fitbit, a kind of accelerometer, provides feedback to subjects combined with an activity counseling program will result in an increase in physical activity of at least 20%.

ELIGIBILITY:
Inclusion criteria

* Volunteers from the public including subjects in the independent living section of Assisted Living Facilities between the ages of 65 and 85.
* Those over 85 may participate with their personal physician's consent.
* BMI 25-40 kg/m2 OR a waist circumference 88 cm or greater in women or 102 cm or greater in men
* Sedentary (no more than 30 minutes of vigorous or 90 minutes of moderate activity per week)
* Complete a Timed Get Up and Go test in <= 20 seconds
* If walking is done with an assistive device, the subject must have no history of falling with the use of said device)
* Subjects will complete the Physical Activity Readiness Questionnaire - Revised (PARQ-R) which is as follows:

  1. Has your doctor ever said that you have a heart condition and that you should only do physical activity recommended by a doctor?
  2. Do you feel pain in your chest when you do physical activity?
  3. In the past month, have you had chest pain when you were not doing physical activity?
  4. Do you lose your balance because of dizziness, or do you ever lose consciousness?
  5. Do you have a bone or joint problem that could be made worse by a change in your physical activity?
  6. Is your doctor currently prescribing drugs (for example, water pills) for your blood pressure or heart condition?
  7. Do you know of any other reason why you should not do physical activity? Subjects who respond "yes" to any of the above questions will require written permission from their physician to participate in this study.

Exclusion criteria:

* Significant cognitive impairment (score on Mini-Cog less than 3).
* Diabetics on medication
* Subjects who should not participate in an exercise program will not be eligible for the study.
* Angina or a history of myocardial infarction
* Cancer (other than non-melanoma skin cancer) will not be eligible.
* Uncompensated liver disease
* Uncompensated thyroid disease
* Severe osteoporosis
* Any medical condition which might lead to weight loss or weight gain
* Patients on the following medications: antidepressants (those on bupropion and stable doses of selective serotonin re-uptake inhibitors (SSRIs) and trazodone will be included), antipsychotics, topiramate, orlistat, or phentermine (Patients on statins will be eligible if no change in their medication is planned over the next 6 months)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Activity units as determined by Accelerometry | 6 and 12 months

SECONDARY OUTCOMES:
Body weight in kilograms | 6 and 12 months
Body fat by bone density scan (DEXA) | 6 and 12 months
Waist to hip ratio | 6 and 12 months
Fasting glucose | 6 and 12 months
Hemoglobin A1c | 6 and 12 months
Fasting insulin | 6 and 12 months
Fasting lipid profile | 6 and 12 months
high sensitivity c-reactive protein | 6 and 12 months
Body Mass Index | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren Thompson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Thompson WG, Kuhle CL, Koepp GA, McCrady-Spitzer SK, Levine JA. "Go4Life" exercise counseling, accelerometer feedback, and activity levels in older people. Arch Gerontol Geriatr. 2014 May-Jun;58(3):314-9. doi: 10.1016/j.archger.2014.01.004. Epub 2014 Jan 15. PMID 24485546